CLINICAL TRIAL: NCT02330835
Title: Multimedia Program to Promote Positive Bus Behavior
Acronym: BUS_2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Lynne Swartz, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR55-2; 1R44DA015251-02 (NIH)
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Student Behavior
Keywords: school; bus; school bus; driver; training; behavior; management; interactive; computer
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In the Driver's Seat (Experimental): Treatment materials. In the Driver's Seat: A Roadmap to Managing Student Behavior on the Bus is a comprehensive multimedia program that guides transportation departments in creating and maintaining a safe, responsible, and positive environment on the school bus through effective student behavior management. The program includes three components: 1) In the Driver's Seat: Transportation Supervisor Program for transportation department administrative staff, 2)In the Driver's Seat: Group Lessons DVD for Drivers. The DVD-based curriculum is designed to be facilitated by a transportation supervisor or driver trainer in groups and 3)In the Driver's Seat: Bus Driver Program. This CD-ROM-based program for bus drivers.
  Interventions: Behavioral: In the Drivers Seat
- School bus driver training videos (Active Comparator): Control materials. Bus drivers in the control condition viewed two linear videos on study computers. In Session 1 of the intervention, Control drivers viewed School Bus Driving, Part 1, 2nd Edition, © 1991, AIMS Media, 23-minute linear video showing defensive driving techniques. In Session 2, Control drivers viewed Decide Smart, Arrive Safe, © 2005, Operation Lifesaver, Inc., a video about school bus safety at railroad crossings produced in conjunction with the National Association of State Directors of Pupil Transportation services. Supervisors in the control condition received no materials until completing the study (waitlisted).
  Interventions: Behavioral: School bus driver training videos

INTERVENTIONS:
Behavioral: In the Drivers Seat — Multimedia student behavior management program for school bus drivers and school administrators
  Other Names: A Roadmap To Managing Student Behavior On the Bus
  Arms: In the Driver's Seat
Behavioral: School bus driver training videos — Basic bus driving safety videos
  Arms: School bus driver training videos

SUMMARY:
This project evaluated a multimedia student behavior management program for school bus drivers and school administrators.

DETAILED DESCRIPTION:
We developed a comprehensive multimedia training program for transportation departments. In the Driver's Seat: A Roadmap to Managing Student Behavior on the Bus guides transportation departments in creating and maintaining a safe, responsible, and positive environment on the bus through drivers' use of effective student behavior management techniques. The program teaches skills for the bus context based on the principles of positive behavior supports and the foundational work of Sprick and colleagues (Sprick, 1990; Sprick, Garrison, & Howard, 2002; Sprick, Sprick, & Garrison, 1992). In the Driver's Seat was designed as a stand-alone DVD-based training program for school bus drivers of elementary schools, using video examples presenting real driver and student interactions on the bus. A computer-based program for transportation supervisors supplemented the driver training materials and included information for supervisors about developing and maintaining department-wide transportation policies, as well as an overview of the bus driver training materials and instructions for their use.

The components of the In the Driver's Seat bus driver training program could be implemented by a transportation team without the need of an expert and could be used to train new personnel or review and refresh veteran personnel's skills. The DVD-based component was designed for use by a transportation supervisor or driver trainer in a group setting with drivers and augmented the material presented in the drivers' program.

ELIGIBILITY:
Inclusion Criteria:

* Bus drivers and administrators will be 18 or older.
* All subjects must be employed by elementary or middle schools.

Exclusion Criteria:

* Excluded from the study will be bus drivers and administrators not in elementary schools
* Staff who are not bus drivers or administrators for elementary or middle schools will also be excluded.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Attitudes and beliefs regarding bus climate | up to 60-day follow up
  The Attitudes and Beliefs regarding Bus Climate items consisted of a total of 27 questions that assessed drivers in the following areas: (1) relationships with students; (2) understanding how to respond to student behavior; (3) interactions with students; (4) drivers' perception of their own bus climate; (5) communication with other drivers; and (6) departmental support for behavior management. For each of the attitudes and beliefs items, drivers were asked how much they agreed, or disagreed, with key statements. For example: "Bus drivers treat students respectfully." The second attitudes/beliefs items assessed drivers' job satisfaction by asking for the driver's level of agreement with statements such as, "I feel like my job is important." Response options were the same for all attitudes/beliefs items: "1=Agree a lot, 5=disagree a lot."

SECONDARY OUTCOMES:
Self-efficacy in managing misbehavior | Session 1 (Day 1) posttest, Session 2 (Day 2) posttest, 30-day follow-up, 60-day follow-p
  Drivers' self-efficacy was assessed by two sets of items. The first set of items assessed drivers' confidence in knowing best ways to deal with misbehaviors. These included 10 items that asked drivers to rate their level of confidence in knowing how to handle specific student misbehaviors such as inappropriate behavior or students physically hurting other students. The second set of items assessed drivers' confidence in using specific strategies. These were four items developed from the program content; e.g., "How confident are you that you could always restate the behavior rule every time a student argues with you?" Each of the self-efficacy items used a 5-point rating scale (1=very confident, 2=somewhat confident, 3=not sure, 4=doubtful, and 5=not at all confident).
Perceived student misbehaviors | Session 1 (Day 1) posttest, Session 2 (Day 2) posttest, 30-day follow-up, 60-day follow-p
  The student misbehaviors items assessed drivers' perception of frequency of student misbehavior occurrences. The items asked drivers to indicate how often student misbehaviors occurred, such as inappropriate language, students damaging or littering the bus, or students threatening or bullying other students. Responses were on a 5-point scale: "1=All of the time, 2=most of the time, 3=about half the time, 4=rarely, and 5=never."
Knowledge | Session 1 (Day 1) posttest, Session 2 (Day 2) posttest, 30-day follow-up, 60-day follow-p
  . Seven knowledge items were developed to test drivers on specific program content from the two main program modules: 1) techniques for creating a positive and safe environment on the bus (i.e., positive environment) and 2) effective strategies for correcting misbehaviors when they occur (i.e., correction strategies). Each item was presented as a multiple-choice question, with 1 correct response and 3 distractors. Each of the 7 items was coded "1" for correct and "0" for incorrect answers. A mean score was then calculated to create a scale.
Intention-behavior | Session 1 (Day 1) posttest, Session 2 (Day 2) posttest, 30-day follow-up, 60-day follow-p
  Items in the intention-behavior scale, adapted from the Parenting Scale by Arnold, O'Leary, Wolff, & Acker (1993),were presented with text anchors on each continuum For example, at the left side of a row of circles a text response represented the more effective response to the student interaction (coded as "7"). At the right side of the row of circles a text response represented the least effective response to the student interaction (coded as "1"). The driver chose the circle corresponding to how he or she would respond. For example, for the statement, "When I correct a student for misbehavior," the response anchors presented were "I state the rule in my correction" (best response; 7 points) and "I say whatever needs to be said without thinking too much about the wording" (least effective response; 1 point). If the driver chose the second circle from the right, the response was coded as a "6." Item scores were summed and a mean score calculated.
Student referrals | Session 1 (Day 1) posttest, Session 2 (Day 2) posttest, 30-day follow-up, 60-day follow-p
  Bus drivers were asked to report the number of referrals they had written within the last 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States

REFERENCES:
- See also: Developer — http://orcasinc.com
- See also: Distributor — http://www.pacificnwpublish.com/